CLINICAL TRIAL: NCT06648616
Title: Evaluating the Effects of Elastic Bands Resistance Training on Performance Parameters in Female Football Players: A Pilot Study
Brief Title: Impact of Elastic Band Resistance Training on Female Football Performance: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Responsible Party: Principal Investigator, Henrique Sousa, Principal Investigator, University of Maia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EBT_HS_01
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Physical Perfrormance Parameters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elastic Band Group (Experimental): Athletes that have participated in a bi-weekly elastic band resistance training program.
  Interventions: Other: EBT

INTERVENTIONS:
Other: EBT — Elastic Band Resistance Training

SUMMARY:
The goal of this clinical trial is to assess the effects of a 6-week strength training program with elastic bands on several physical components in adult female football players. The main question it aims to answer is:

Will a specific elastic band resistance training help improve some components of physical performance in adult female football players?

Participants will perform a bi-weekly elastic band resistance training, during a period of 6-weeks. This program will be incorporated into their in-season regimen, before their training session.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years of age;
* belong in the senior level of an amateur or professional women´s football club;
* play in one of the three Portuguese national women´s football leagues.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Knee extension and flexion isometric strength | At the beginning and end of the study (Week 1 and Week 6)
  Maximal isometric knee extension and flexion force will be measured using a handheld dynamometer (DynaMo Plus, VALD Performance, Brisbane, Queensland, Australia). For the knee extension assessment, participants will be in a seated position, whereas during the knee flexion evaluation, the participants will be in a prone position. To generate their maximal torque, the dynamometer chain length will be adjusted so that their knee angle will be at ∼60° and ∼30°, for the knee extension and flexion, respectively. Participants will then apply a maximal isometric effort, maintaining it for 5s, without any subsidiary body movements.
Vertical jump | At the beginning and end of the study (Week 1 and Week 6)
  Jump height was evaluated using an optical measurement system (OptoJump, Microgate, Bolzano, Italy). The players will perform the countermovement jump, where they will begin from an upright position; a rapid downward movement to a knee angle of ∼90°, immediately transitioning to propel themselves upwards into the air.
Change of direction sprint | At the beginning and end of the study (Week 1 and Week 6)
  The Modified T-Test will be implemented to assess change of direction sprint. This evaluation has within itself directional changes such as forward sprinting, left and right-side shuffling, and backpedaling. Photocells (WhittyGate, Microgate, Bolzano, Italy) will be used for a more precise time count.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maia, Maia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided